CLINICAL TRIAL: NCT06557356
Title: A Dose-Escalation Phase 1, Investigator- and Participant-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of LY3532226 in Participants With Obesity
Brief Title: A Study of LY3532226 in Participants With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18835; J2V-MC-GZLD (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3532226 (Part A) (Experimental): LY3532226 administered subcutaneously (SC)
  Interventions: Drug: LY3532226
- Placebo (Part A) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- LY3532226 (Part B) (Experimental): LY3532226 administered SC
  Interventions: Drug: LY3532226
- Placebo (Part B) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo
- LY3532226 (Part C) (Experimental): LY3532226 administered SC
  Interventions: Drug: LY3532226
- Placebo (Part C) (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3532226 — Administered SC
  Arms: LY3532226 (Part A); LY3532226 (Part B); LY3532226 (Part C)
Drug: Placebo — Administered SC
  Arms: Placebo (Part A); Placebo (Part B); Placebo (Part C)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug known as LY3532226 in participants with obesity. Blood tests will be performed to check how much LY3532226 gets into the bloodstream and how long it takes the body to eliminate it following weekly or monthly administration. Part A of the study will last approximately 16 weeks, excluding screening period. Part B of the study will last approximately 20 weeks, excluding the screening period. Part C of the study will last approximately 8 weeks, excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have a body weight not exceeding 150 kilograms (kg) or 330 pounds (lb) and body mass index (BMI) within the range of 30 to 40 kilogram per square meter (kg/m²)
* Have had a stable body weight that is less than or equal to 5% change in body weight for 3 months prior to screening and enrollment

Exclusion Criteria:

* Have a lifetime history of a suicide attempt
* Have a history or presence of psychiatric disorders, including a history of major depressive disorder within the last 2 years
* Have a baseline Patient Health Questionnaire-9 (PHQ-9) score of 15 or greater, and/or a score of 2 or greater for either of the first 2 questions on the PHQ-9 questionnaire
* Have a known clinically significant gastric emptying abnormality, have undergone gastric bypass surgery or restrictive bariatric surgery
* Have taken approved or investigational medication for weight loss, within the previous 3 months or 5 half-lives of study screening, whichever is earlier
* Intend to use any weight-loss medications during study participation
* Have obesity induced by other endocrinologic disorders or diagnosed monogenetic or syndromic forms of obesity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 16 Weeks)
  A summary of TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module
Part B: Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 20 Weeks)
  A summary of TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module
Part C: Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 8 Weeks)]
  A summary of TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Part A: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3532226 | Predose on Day 1 through Week 16
  PK: Cmax of LY3532226
Part A: PK: Area Under the Concentration Versus Time Curve (AUC) of LY3532226 | Predose on Day 1 through Week 16
  PK: AUC of LY3532226
Part B: PK: Cmax of LY3532226 | Predose on Day 1 through Week 20
  PK: Cmax of LY3532226
Part B: PK: AUC of LY3532226 | Predose on Day 1 through Week 20
  PK: AUC of LY3532226
Part C: Pharmacodynamic (PD): Change in insulin sensitivity index (Si) | Baseline up to Approximately Week 4
  Part C: PD: Change in Si

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (3):
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Fortrea Clinical Research Unit, Dallas, Texas
  - Fortrea Clinical Research Unit, Madison, Wisconsin
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lilly Trials — https://trials.lilly.com/en-US/trial/527756